CLINICAL TRIAL: NCT03259399
Title: A Study of Genetic Variants Associated With Enalapril-Induced Adverse Drug Reaction and Impact of Pharmacogenomics on First Stroke in Hypertensive Patients Taking Enalapril or Enalapril-Folic Acid Therapy.
Brief Title: A Pharmacogenomics Study of Safety and Efficacy of Enalapril or Enalapril-Folic Acid Therapy in Hypertensive Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cui Yimin (Other)
Responsible Party: Sponsor-Investigator, Cui Yimin, Director of pharmacy，M.D & Ph.D, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: 2016[1238]
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Enalapril Adverse Reaction; Pharmacogenomics; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- wild genotype: Detection of genotype will be carried out through next generation sequencing, distinguish wild genotype of enalapril
  Interventions: Genetic: detection of genotype
- mutant genotype: Detection of genotype will be carried out through next generation sequencing, distinguish mutant genotype of enalapril
  Interventions: Genetic: detection of genotype

INTERVENTIONS:
Genetic: detection of genotype — detection of genotype by next generation sequencing

SUMMARY:
Dry cough is the most common adverse reaction of angiotensin converting enzyme, including enalapril, in Chinese population. Clinical observations suggest that the incidence of ACEI-induced dry cough is different between Chinese and other racial groups, however, there is still lack of research data in Chinese. Stroke is the second leading cause of death in the world and leading cause of death in China. Except the known risk factor such as hypertension, high homocysteine level, folic acid deficiency, the impact of genetics should not be ignored.

In this study, we will investigate whether there are specific genotypes which may predict the incidence of (1)enalapril-induced dry cough in Chinese and (2)first stroke in hypertensive patients taking enalapril or enalapril-folic acid therapy, so as to provide a basis for developing guidelines on precision medication in enalapril therapy apply to Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Patients taking enalapril or enalapril-folic acid therapy
* Signed informed consent.

Exclusion Criteria:

* Patients not taking enalapril treated
* Intolerance or unwillingness to blood sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Patients:In accordance with anti-hypertension indications of enalapril
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2017-08-16 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dry cough | At 2 years
First Incidence of stroke | At 2 years

SECONDARY OUTCOMES:
Genotype detected by next generation sequencing | pre-dose of enalapril or enalapril-folic acid (Baseline)
  Collect blood specimen before enalapril administration, then detect genotype of enalapril by next generation sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Mu G, Xie Q, Liu Z, Zhang H, Meng X, Song J, Zhou S, Wang Z, Wang Z, Zhao X, Jiang J, Liao M, Bao J, Zhang F, Xiang Q, Cui Y. Identification of genetic biomarkers associated with pharmacokinetics and pharmacodynamics of apixaban in Chinese healthy volunteers. Expert Opin Drug Metab Toxicol. 2023 Jan;19(1):43-51. doi: 10.1080/17425255.2023.2184344. Epub 2023 Mar 3. PMID 36867504
- [Derived] Mu G, Xiang Q, Zhang Z, Liu C, Zhang H, Liu Z, Pang X, Jiang J, Xie Q, Zhou S, Wang Z, Hu K, Wang Z, Jiang S, Qin X, Cui Y. PNPT1 and PCGF3 variants associated with angiotensin-converting enzyme inhibitor-induced cough: a nested case-control genome-wide study. Pharmacogenomics. 2020 Jun;21(9):601-614. doi: 10.2217/pgs-2019-0167. Epub 2020 May 13. PMID 32397904